CLINICAL TRIAL: NCT01323959
Title: Evaluation of GSK Biologicals' Boostrix™ Polio in Healthy Adults, 10 Years After a Booster Vaccination
Brief Title: Immunogenicity and Safety of Booster Dose of BoostrixTM Polio Vaccine in Previously Boosted Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113060
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-04

CONDITIONS: Acellular Pertussis; Poliomyelitis; Diphtheria; Tetanus
Keywords: BoostrixTM Polio; dTpa-IPV; booster
MeSH Terms: conditions — Poliomyelitis; Diphtheria; Tetanus

ARMS (3):
- BOOSTRIX POLIO GROUP (Experimental): Healthy subjects who had received one booster dose Boostrix™ Polio vaccine in the NCT01277705 study received one additional booster dose of Boostrix™ Polio vaccine in this study, administered as an intramuscular injection into the deltoid region of the left arm.
  Interventions: Biological: BoostrixTM Polio
- BOOSTRIX+POLIORIX GROUP (Experimental): Healthy subjects who had received one booster dose of the co-administered Boostrix™ and Poliorix™ vaccines in the NCT01277705 study received one booster dose Boostrix™ Polio vaccine in this study, administered as an intramuscular injection into the deltoid region of the left arm.
  Interventions: Biological: BoostrixTM Polio
- REVAXIS GROUP (Experimental): Healthy subjects who had received one booster dose of Revaxis® vaccine in the NCT01277705 study received one booster dose of Boostrix™ Polio vaccine in this study, administered as an intramuscular injection into the deltoid region of the left arm.
  Interventions: Biological: BoostrixTM Polio

INTERVENTIONS:
Biological: BoostrixTM Polio — Single dose, intramuscular administration.

SUMMARY:
This study will evaluate the persistence of immune response against diphtheria, tetanus, pertussis and poliomyelitis in healthy adults, 10 years after a booster dose, and also assess the immunogenicity and safety of another booster dose of BoostrixTM Polio.

DETAILED DESCRIPTION:
This protocol posting has been updated following protocol amendment 1, dated 03 June 2011. The impacted section is: Eligibility Criteria (Exclusion criteria).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Male or female subjects who have received vaccine in study NCT01277705.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study and receive the booster vaccine, if the subject:

  * practices/has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * agrees to continue adequate contraception during the entire booster epoch.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the booster dose of the study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the booster dose.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to booster vaccination, or planned administration during the active study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Previous booster vaccination against diphtheria, tetanus, pertussis or poliovirus since the dose received in study NCT01277705. In Germany, previous dose of a monovalent vaccine against pertussis is allowed for subjects in the Group C.
* History of diphtheria, tetanus, pertussis or poliomyelitis diseases following the receipt of booster dose in study NCT01277705.
* Any confirmed or suspected immunosuppressive or immunodeficiency condition based on medical history and physical examination.
* Occurrence of transient thrombocytopenia or neurological complications following an earlier immunisation against diphtheria and/or tetanus.
* Occurrence of any of the following adverse event after a previous administration of a DTP vaccine:

  * Hypersensitivity reaction to any component of the vaccine,
  * encephalopathy of unknown aetiology occurring within seven days following previous vaccination with pertussis-containing vaccine,
  * fever ≥ 40°C within 48 hours of vaccination not due to another identifiable cause,
  * collapse or shock-like state within 48 hours of vaccination,
  * convulsions with or without fever, occurring within 3 days of vaccination.
* Administration of immunoglobulins and/or any blood products within the three months preceding the booster dose or planned administration during the study period.
* Acute disease and/or fever at the time of enrolment.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2011-04-01; Primary Completion 2012-03-01 (Actual); Study Completion 2012-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- France (5):
  - GSK Investigational Site, Derval
  - GSK Investigational Site, La Chapelle-Basse-Mer
  - GSK Investigational Site, La Riche
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Tours
- Germany (8):
  - GSK Investigational Site, Deggendorf, Bavaria
  - GSK Investigational Site, Höhenkirchen-Siegertsbrunn, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Selbitz, Bavaria
  - GSK Investigational Site, Vilshofen, Bavaria
  - GSK Investigational Site, Weilheim, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Kovac M, Rathi N, Kuriyakose S, Hardt K, Schwarz TF. Immunogenicity and reactogenicity of a decennial booster dose of a combined reduced-antigen-content diphtheria-tetanus-acellular pertussis and inactivated poliovirus booster vaccine (dTpa-IPV) in healthy adults. Vaccine. 2015 May 21;33(22):2594-601. doi: 10.1016/j.vaccine.2015.03.104. Epub 2015 Apr 14. PMID 25882172
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 113060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 212 subjects enrolled, 1 subject number was allocated without the study vaccine being administered to that subject, therefore the total number of subjects was 211.
Period: Overall Study
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Started | 67 | 72 | 72
Completed | 67 | 72 | 72
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group | Total
Number analyzed (Participants) | 67 | 72 | 72 | 211
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.4 (12.82) | 49.2 (12.53) | 51.4 (13.06) | 50.33 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 47 | 39 | 121
  Male | 32 | 25 | 33 | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Diphteria (D) and Tetanus (T) Antigens
Description: A seroprotected subject is defined as a vaccinated subject with anti-D and anti-T antibody concentration greater than or equal to (≥) 0.1 international units per millilitre (IU/mL).
Time Frame: At Month 1
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included subjects who met all eligibility criteria, complied with the procedures defined in the protocol, who received the booster dose of Boostrix™ Polio vaccine and for whom data concerning immunogenicity outcome measures were available.
Measure: Number; unit: Subjects
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 63 | 69 | 69
Subjects
  Anti-D | 61 | 66 | 68
  Anti-T | 63 | 69 | 69
Statistical Analysis 1: Comparison: Boostrix Polio Group; The objective of the analysis was to demonstrate that a booster dose of Boostrix™ Polio vaccine, administered to adults 10 years after a dose of Boostrix™ Polio vaccine or co-administered Boostrix™ + Poliorix™ vaccines, elicited seroprotective antibody concentrations, 1 month after the booster dose, in at least 80% of the subjects against diphtheria. Samples were analysed both with ELISA (enzyme-linked immunosorbent assay), and VERO-cell (African green monkey kidney cell) neutralisation testing; Test type: Superiority or Other; Percentage of subjects seroprotected = 96.8, 95% CI 2-sided [89 to 99.6] — The pre-specified lower limit (LL) of the 95% confidence interval (CI) for the percentage of seroprotected (Anti-D concentrations ≥ 0.1 IU/mL by ELISA or ≥ 0.01 IU/mL by VERO-cell when subjects with ELISA result <0.1 IU/mL) subjects was above 80%
Statistical Analysis 2: Comparison: Boostrix+Poliorix Group; The objective of the analysis was to demonstrate that a booster dose of Boostrix™ Polio vaccine, administered to adults 10 years after a dose of Boostrix™ Polio vaccine or co-administered Boostrix™ + Poliorix™ vaccines, elicited seroprotective antibody concentrations, one month after the booster dose, in at least 80% of the subjects against diphtheria; Test type: Superiority or Other; Percentage of subjects seroprotected = 95.7, 95% CI 2-sided [87.8 to 99.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Revaxis Group; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Percentage of subjects seroprotected = 100, 95% CI 2-sided [94.8 to 100] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Number of Seroprotected Subjects Against Poliovirus Types 1, 2 and 3
Description: A seroprotected subject is defined as a vaccinated subject with anti-poliovirus types 1, 2 and 3 antibody concentration greater than or equal to (≥) 8 Effective Dose 50 (ED50)
Time Frame: At Month 1
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 58 | 62 | 60
Subjects
  Anti-polio 1: number analyzed (Participants) | 58 | 62 | 59
  Anti-polio 1 | 58 | 62 | 58
  Anti-polio 2: number analyzed (Participants) | 46 | 58 | 56
  Anti-polio 2 | 46 | 58 | 56
  Anti-polio 3: number analyzed (Participants) | 58 | 60 | 60
  Anti-polio 3 | 58 | 60 | 60

3. Primary Outcome: Number of Seroprotected Subjects Against Diphteria (D) and Tetanus (T) Antigens
Description: as for outcome 1
Time Frame: At Day 0
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 63 | 69 | 69
Subjects
  Anti-D: number analyzed (Participants) | 63 | 68 | 69
  Anti-D | 51 | 50 | 55
  Anti-T | 62 | 68 | 65
Statistical Analysis 1: Comparison: Boostrix Polio Group; The objective of the analysis was to dose in study NCT01277705. Samples were analysed both with ELISA (enzyme-linked immunosorbent assay), and VERO-cell (African green monkey kidney cell) neutralisation testing; Test type: Superiority or Other; Percentage of subjects seroprotected = 92.1, 95% CI 2-sided [82.4 to 97.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Boostrix+Poliorix Group; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Percentage of subjects seroprotected = 79.4, 95% CI 2-sided [67.9 to 88.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Revaxis Group; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Percentage of subjects seroprotected = 84.1, 95% CI 2-sided [73.3 to 91.8] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Number of Seroprotected Subjects Against Poliovirus Types 1, 2 and 3
Description: as for outcome 2
Time Frame: At Day 0
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 58 | 66 | 67
Subjects
  Anti-polio 1: number analyzed (Participants) | 52 | 58 | 60
  Anti-polio 1 | 52 | 58 | 59
  Anti-polio 2: number analyzed (Participants) | 56 | 60 | 63
  Anti-polio 2 | 56 | 60 | 62
  Anti-polio 3 | 57 | 65 | 67

5. Primary Outcome: Number of Subjects With Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA), Anti-pertactin (Anti-PRN) Antibodies
Description: Cut-off values assessed were greater than or equal to ≥ 5 Enzyme Linked Immunosorbent Assay (ELISA) units per millilitre (EL.U/ml)
Time Frame: At Day 0
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 62 | 69 | 69
Subjects
  Anti-PT: number analyzed (Participants) | 61 | 69 | 69
  Anti-PT | 48 | 58 | 49
  Anti-FHA: number analyzed (Participants) | 62 | 69 | 67
  Anti-FHA | 62 | 69 | 66
  Anti-PRN: number analyzed (Participants) | 62 | 68 | 69
  Anti-PRN | 55 | 64 | 59

6. Primary Outcome: Anti-diphteria (Anti-D) and Anti-tetanus (Anti-T) Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in international units per millilitre (IU/mL)
Time Frame: At Day 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 63 | 69 | 69
IU/mL
  Anti-D: number analyzed (Participants) | 63 | 68 | 69
  Anti-D | 0.416 [0.293 to 0.592] | 0.360 [0.249 to 0.519] | 0.501 [0.348 to 0.721]
  Anti-T | 1.371 [1.019 to 1.844] | 1.578 [1.227 to 2.028] | 1.491 [1.096 to 2.028]

7. Primary Outcome: Anti-polio 1, Anti-polio 2 and Anti-polio 3 Antibody Titers
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: At Day 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 58 | 66 | 67
Titers
  Anti-polio 1: number analyzed (Participants) | 52 | 58 | 60
  Anti-polio 1 | 341.0 [233.5 to 497.9] | 567.0 [392.3 to 819.4] | 332.0 [239.0 to 461.2]
  Anti-polio 2: number analyzed (Participants) | 56 | 60 | 63
  Anti-polio 2 | 308.3 [218.9 to 434.3] | 322.6 [234.3 to 444.2] | 331.5 [246.3 to 446.0]
  Anti-polio 3 | 388.9 [271.2 to 557.7] | 648.5 [476.7 to 882.2] | 542.1 [397.1 to 740.1]

8. Primary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA), Anti-pertactin (Anti-PRN) Antibodies Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in expressed in ELISA units per millilitre (EL.U/mL)
Time Frame: At Day 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 62 | 69 | 69
EL.U/mL
  Anti-PT: number analyzed (Participants) | 61 | 69 | 69
  Anti-PT | 10.3 [8.2 to 13] | 13.4 [10.4 to 17.2] | 14.7 [10.1 to 21.5]
  Anti-FHA: number analyzed (Participants) | 62 | 69 | 67
  Anti-FHA | 93.7 [72.9 to 120.6] | 124.0 [102.5 to 150.1] | 68.6 [49.2 to 95.9]
  Anti-PRN | 66.1 [41.9 to 104.1] | 93.9 [62.7 to 140.7] | 19.4 [14.2 to 26.5]

9. Secondary Outcome: Number of Subjects With Booster Response to Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA), Pertactin (PRN)
Description: Booster response was defined as: for initially seronegative subjects: antibody concentration ≥ 20 EL.U/mL at post booster vaccination; for initially seropositive subjects with pre-vaccination antibody concentration < 20 EL.U/mL: antibody concentration at post booster ≥ 4 fold the pre-vaccination antibody concentration; and for initially seropositive subjects with pre-vaccination antibody concentration ≥ 20 EL.U/mL: antibody concentration at post booster ≥ 2 fold the pre-vaccination antibody concentration.
Time Frame: At Month 1
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 62 | 69 | 69
Subjects
  Anti-PT: number analyzed (Participants) | 61 | 69 | 68
  Anti-PT | 60 | 60 | 52
  Anti-FHA: number analyzed (Participants) | 62 | 69 | 67
  Anti-FHA | 53 | 62 | 57
  Anti-PRN: number analyzed (Participants) | 62 | 68 | 69
  Anti-PRN | 46 | 43 | 63

10. Secondary Outcome: Number of Subjects With Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA), Anti-pertactin (Anti-PRN) Antibodies Above the Cut-off
Description: as for outcome 5
Time Frame: At Month 1
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 63 | 69 | 69
Subjects
  Anti-PT: number analyzed (Participants) | 63 | 69 | 68
  Anti-PT | 63 | 69 | 67
  Anti-FHA | 63 | 69 | 69
  Anti-PRN | 63 | 69 | 69

11. Secondary Outcome: Anti-diphteria (Anti-D) and Anti-tetanus (Anti-T) Antibody Concentrations
Description: as for outcome 6
Time Frame: At Month 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 63 | 69 | 69
IU/mL
  Anti-D | 2.159 [1.579 to 2.952] | 1.821 [1.312 to 2.528] | 2.649 [1.948 to 3.603]
  Anti-T | 8.568 [7.361 to 9.972] | 9.692 [8.217 to 11.431] | 9.390 [7.946 to 11.096]

12. Secondary Outcome: Anti-polio 1, Anti-polio 2 and Anti-polio 3 Antibody Titers
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: At Month 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 58 | 62 | 60
Titers
  Anti-polio 1: number analyzed (Participants) | 58 | 62 | 59
  Anti-polio 1 | 1519.0 [1156.9 to 1994.4] | 1665.4 [1263.5 to 2195.2] | 1526.7 [1106.8 to 2105.9]
  Anti-polio 2: number analyzed (Participants) | 46 | 58 | 56
  Anti-polio 2 | 1071.3 [806.2 to 1423.5] | 1269.8 [954.5 to 1689.4] | 1550.1 [1202.8 to 1997.7]
  Anti-polio 3: number analyzed (Participants) | 58 | 60 | 60
  Anti-polio 3 | 2035.7 [1653.4 to 2506.4] | 2047.9 [1604.6 to 2613.7] | 2024.6 [1513.3 to 2708.6]

13. Secondary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA), Anti-pertactin (Anti-PRN) Antibodies Antibody Concentrations
Description: as for outcome 8
Time Frame: At Month 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 63 | 69 | 69
EL.U/mL
  Anti-PT: number analyzed (Participants) | 63 | 69 | 68
  Anti-PT | 97.5 [81.4 to 116.9] | 100.1 [80.3 to 124.8] | 92.9 [68.7 to 125.6]
  Anti-FHA | 485.8 [413.8 to 570.4] | 553.5 [465.9 to 657.6] | 854.9 [714.9 to 1022.3]
  Anti-PRN | 365.9 [281.5 to 475.6] | 404.2 [324.2 to 504.0] | 581.0 [401.6 to 840.7]

14. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 4-day (Day 0-Day 3) follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with documented administration of the study booster vaccine, for whom data was available.
Measure: Number; unit: Subjects
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 67 | 72 | 72
Subjects
  Pain, Any | 42 | 49 | 46
  Pain, Grade 3 | 0 | 0 | 0
  Rednes, Any | 22 | 26 | 32
  Redness, >50 mm | 1 | 4 | 3
  Swelling, Any | 18 | 21 | 19
  Swelling, >50 mm | 0 | 3 | 1

15. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Assessed solicited general symptoms were fatigue, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], headache and gastrointestinal symptoms. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Day 0-Day 3) follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with documented administration of the study booster vaccine, for whom data was available and the symptom sheet filled in.
Measure: Number; unit: Subjects
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 65 | 71 | 71
Subjects
  Fatigue, Any | 12 | 16 | 15
  Fatigue, Grade 3 | 1 | 1 | 0
  Fatigue, Related | 9 | 11 | 9
  Gastrointestinal symptoms, Any | 7 | 9 | 4
  Gastrointestinal symptoms, Grade 3 | 0 | 0 | 0
  Gastrointestinal symptoms, Related | 3 | 4 | 3
  Headache, Any | 7 | 11 | 11
  Headache, Grade 3 | 0 | 0 | 0
  Headache, Related | 6 | 6 | 9
  Fever (axillary), ≥ 37.5 °C | 3 | 2 | 1
  Fever (axillary), > 39 °C | 0 | 0 | 0
  Fever (axillary), Related | 1 | 2 | 1

16. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs).
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Day 0-Day 30) follow-up period after vaccination
Population: as for outcome 15
Measure: Number; unit: Subjects
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 67 | 72 | 72
Subjects | 6 | 5 | 6

17. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Month 0 - Month 1
Population: as for outcome 14
Measure: Number; unit: Subjects
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Number analyzed (Participants) | 67 | 72 | 72
Subjects | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms during the 4-day post-vaccination period (Days 0-3), Unsolicited AEs during the 31-day post-vaccination (Days 0-30), SAEs during the entire study period (Month 0 - 1).
Arm/Group | Boostrix Polio Group | Boostrix+Poliorix Group | Revaxis Group
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 52/67 | 54/72 | 54/72
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Boostrix Polio Group (N=67) | Boostrix+Poliorix Group (N=72) | Revaxis Group (N=72)
Pain (General disorders) | 42 | 49 | 46
Redness (General disorders) | 22 | 26 | 32
Swelling (General disorders) | 18 | 21 | 19
Fatigue (General disorders) | 12/65 | 16/71 | 15/71
Gastrointestinal symptom (General disorders) | 7/65 | 9/71 | 4/71
Headache (General disorders) | 7/65 | 11/71 | 11/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.